CLINICAL TRIAL: NCT06889935
Title: The Effect of Respiratory Exercise Diary Use on Postoperative Pain in Patients Undergoing Cardiovascular Surgery
Brief Title: Investigating the Effect of Respiratory Exercise Diary on Pain in Cardiovascular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Melisa Köse, Principal Investigator, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MARU-SBF-MKT-01
Record Dates: First submitted 2025-03-16; First posted 2025-03-21 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Surgery
Keywords: Cardiovascular surgery; exercise diary; nursing care; pain; postoperative pain; postoperative period; respiratory exercise; spirometer
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Two groups with a conventional therapy control group
Who Masked: Participant, Outcomes Assessor
Masking Description: In order to avoid bias in the people included in the study, randomisation was performed. The randomisation table was created by using the address 'https://www.calculatorsoup.com'.
  In this study, full (double) blinding was not possible because the researcher was the one who implemented the intervention. However, since the participants did not know which group they were included in, blinding was provided at the level of the participants. Blinding was performed while obtaining 'Informed Voluntary Consent'. In this study, in which single blinding method was used, an external biostatistician was assigned during the statistical analysis process and thus blinding was also performed at the analysis stage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group using a respiratory exercise diary (intervention group) (Active Comparator): All of the patients included in the group were asked to fill in the 'Patient Identification Form' and pain assessment was performed with 'Visual Analogue Scale (VAS)'. Information was given about respiratory exercises and spirometry, which is routinely used in the postoperative period in patients undergoing cardiovascular surgery in the hospital where the study was conducted. Respiratory Exercise Diary was introduced to this group and its use was demonstrated practically. They were asked to record the exercises performed in this diary. Pain assessment was performed with Visual Analogue Scale for the first 3 days after surgery. On the 1st postoperative day, this group was informed again about respiratory exercises, spirometer and its daily use, and the first exercises and records were made together with the researcher. They were asked to continue the exercises and recordings themselves for the first 3 days.
  Interventions: Other: Exercise diary
- Group not using a respiratory exercise diary (control group) (No Intervention): 'Patient Identification Form' was filled out for all patients and pain assessment was performed with 'Visual Analogue Scale (VAS)'. Information was given about respiratory exercises and spirometry, which is routinely used in the postoperative period in patients undergoing cardiovascular surgery in the hospital where the study was conducted. This group was asked to note the exercises on a piece of paper. Pain assessment was performed with Visual Analogue Scale in the first 3 days postoperatively. On the 1st postoperative day, the information about breathing exercises and recording procedures was repeated and the practices continued in the routine functioning of the clinic.

INTERVENTIONS:
Other: Exercise diary — The respiratory exercise diary was prepared by reviewing the literature in order to record the time, number and frequency of respiratory exercises performed by patients with the use of a spirometer. On the first page of the diary consisting of two pages; the patient's name and surname, date of surgery, date of birth, how and how often to use the spirometer, and a pictorial information note to remind the position to be taken were included, while on the second page; the chart in which the patients would write the number of exercises they performed with the spirometer during the first three postoperative days opposite the relevant hour was included.
  Other Names: Respiratory exercise diary
  Arms: Group using a respiratory exercise diary (intervention group)

SUMMARY:
The study was carried out to evaluate the effect of respiratory exercise diary use on postoperative pain in patients undergoing elective cardiovascular surgery in a training and research hospital in Istanbul.

DETAILED DESCRIPTION:
The randomised controlled experimental study was conducted between 11 July 2024 and 11 January 2025 in the cardiovascular surgery inpatient wards of a training and research hospital in Istanbul. The study was conducted with a total of 74 patients, 37 in the control group and 37 in the intervention group. Data were collected by the researcher through face-to-face interviews with the patients. 'Patient Identification Form', "Visual Analogue Scale (VAS)", "Respiratory Exercise Diary" were used.

ELIGIBILITY:
Inclusion Criteria:

* No barriers to verbal communication (mental, physiological and psychological)
* Patients undergoing elective cardiovascular surgery,
* Individuals who agreed to participate in the study,
* Patients whose haemodynamics are suitable for respiratory exercise

Exclusion Criteria:

* Being in the intensive care unit after surgical intervention,
* Patients undergoing re-operation after surgical intervention,
* Those who do not accept the study or who want to leave during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2025-01-11 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | four days
  VAS is a very common scale used for pain assessment in daily practice and in this assessment, pain averages ranging from 0 to 10 are given on a 10 cm straight line in a horizontal or vertical plane. In the scale used to determine the pain intensity of patients, pain is graded between 0 (no pain) and 10 (unbearable pain). Accordingly, while '0' indicates no pain, an average VAS value of less than 3 indicates mild pain, 3-6 indicates mild-moderate pain, and greater than 6 indicates moderate-severe pain. VAS is an accepted scale in the world literature that visually describes pain intensity, provides ease of use and consists of a single question.

CONTACTS AND LOCATIONS:
Overall Officials: Melisa KÖSE TUNÇ, Student, Principal Investigator — Marmara University; Hamdiye B. KATRAN, Asst. Prof., Principal Investigator — Marmara University; Mehmet E. MEMETOĞLU, Assoc. Prof., Principal Investigator — Dr. Siyami Ersek Training and Research Hospital Department of Cardiovascular Surgery
Locations (1):
- Marmara Univesity, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No